CLINICAL TRIAL: NCT05106205
Title: An Open Label, Randomized, Single Dose, Crossover Study to Evaluate the Pharmacokinetics and Safety of DA-5213 10mg in Healthy Subjects
Brief Title: Phamacokinetics and Safety Profiles of DA-5213 10mg in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIBE2021-55
Record Dates: First submitted 2021-10-24; First posted 2021-11-03 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental)
  Interventions: Drug: DA-5213 10mg; Drug: DA-5213-R 10mg
- Sequence B (Experimental)
  Interventions: Drug: DA-5213 10mg; Drug: DA-5213-R 10mg

INTERVENTIONS:
Drug: DA-5213 10mg — single dose administration (one tablet once a day)
Drug: DA-5213-R 10mg — single dose administration (one tablet once a day)

SUMMARY:
Phamacokinetics and safety profiles of DA-5213 10mg in Healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* BMI between 18.0 and 30.0 kg/m2
* Body weight : Male≥50kg, Female≥45kg

Exclusion Criteria:

* Allergy or Drug hypersensitivity
* Clinically significant Medical History

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
AUCt | [Time Frame: pre-dose~48 hours post-dose]
  area under the curve
Cmax | [Time Frame: pre-dose~48 hours post-dose]
  maximum plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital, Siheung-si, Gyeonggi-do, South Korea